CLINICAL TRIAL: NCT01255228
Title: Effect of Low Glycemic Index Diet on Body Composition and Mechanism of Obese
Brief Title: Effect of Low Glycemic Index Diet on Body Composition and Mechanism of Obese Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Jen-Fang Liu, Taipei Medical University, School of Nutrition and Health Sciences
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 99055
Record Dates: First submitted 2010-11-18; First posted 2010-12-07 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-12

CONDITIONS: Obesity
Keywords: obesity; body composition; adipocyte-derived cytokine; low glycemic index
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low glycemic index diet (Experimental): The study expect that long-term low GI diet intervention have beneficial effects on regulate body composition of obese women
  Interventions: Other: Low glycemic index diet
- diet intervention (Experimental): The study expect that long-term low GI diet intervention have beneficial effects on regulate body composition of obese women
  Interventions: Other: Low glycemic index diet

INTERVENTIONS:
Other: Low glycemic index diet — The study expect that long-term low GI diet intervention have beneficial effects on regulate body composition of obese women

SUMMARY:
Excessive body weight and obesity have reached epidemic proportions over the last few decades, which may cause many chronic diseases. Maintaining a healthy life style could decrease the risk for obesity, metabolic syndrome and cardiovascular disease. The study aimed to evaluate long-term low glycemic index (GI) diet intervention on lipid profile, body composition and the mechanism of obese women. The pilot study will recruit twenty healthy subjects, and served test food to determine low GI food. In the experiment period, twenty women age from 20-50 years will be recruited. To be included in the study, subjects should have a BMI above 24 kg/m2, or the either one (fat mass ≧ 30% or waistline > 80 cm). Before dietary intervention, participants will receive food choice table and dietary questionnaires to record their dietary intake.

The study will be a randomized, crossover, controlled clinical trails. The experiment period have six weeks, each participants will provide low GI diet (lunch and dinner). On the 0, 3, 6 week, subjects will measurement their body composition (body weight, body mass, waist and hip circumferences) and collect fasting blood samples to analysis the lipid profile, free fatty acid, blood sugar, insulin, adiponectin, leptin and fatty acid synthesis enzymes. Statistical analysis will be performed by paired t-test. The study expect that long-term low GI diet intervention have beneficial effects on regulate body composition of obese women.

ELIGIBILITY:
Inclusion Criteria:

* BMI above 24 kg/m2, or the either one ( fat mass ≧ 30% or waistline > 80 cm )

Exclusion Criteria:

* Cardiovascular disease
* type 2 diabetes mellitus or impaired glucose tolerance
* serious liver or renal disease, gastro-intestinal disease
* proceed serious diet control for formerly three months
* take any supplemental food products or medications known to influence lipid or carbohydrate metabolism

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-02 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
the effect of body composition ( body weight,body mass,waist and hip circumferences ) | 6 week

CONTACTS AND LOCATIONS:
Overall Officials: Jen-Fang Liu, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan